CLINICAL TRIAL: NCT03559114
Title: PROTEST Trial - PROphylaxis for Venous ThromboEmbolism in Severe Traumatic Brain Injury, a Double-blind Randomized Controlled Trial
Brief Title: PROphylaxis for Venous ThromboEmbolism in Severe Traumatic Brain Injury (PROTEST)
Acronym: PROTEST
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Sunnybrook Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 0785
Record Dates: First submitted 2018-04-10; First posted 2018-06-15 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: Traumatic Brain Injury
Keywords: Sequential Compression Device; Anticoagulant Thromboprophylaxis; Deep Vein Thrombosis; Sub Cutaneous; VTE
MeSH Terms: conditions — Brain Injuries, Traumatic; Venous Thrombosis | interventions — Dalteparin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Anticoagulant (Active Comparator): Dalteparin sodium (at a dose of 5000 IU once daily by subcutaneous injection) for 7 days upon randomization after hospital admission.
  Interventions: Drug: Dalteparin
- Saline (Placebo Comparator): Saline (0.2 mL) once daily by subcutaneous injection for 7 days upon randomization after hospital admission.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Dalteparin — Dalteparin in prophylactic doses administered daily if screening criteria are satisfied.
  Other Names: Fragmin
  Arms: Anticoagulant
Drug: Saline — Saline in prophylactic doses administered daily if screening criteria are satisfied.
  Other Names: Sodium Chloride
  Arms: Saline

SUMMARY:
This is a phase III, multi-centre, double blind, randomized controlled trial of patients with traumatic brain injury (TBI).

DETAILED DESCRIPTION:
Patients with severe brain injury are at risk for developing blood clots in their legs, which can travel to the lungs. This potentially serious complication is known as venous thromboembolism (VTE). Anticoagulants are commonly used to prevent VTE in hospital patients. However, in patients with major head injury, anticoagulant prevention is commonly delayed for the fear that it can potentially lead to further bleeding in the brain. Another method that aims to prevent blood clots involves the use of sequential compression device (SCD) that compress the legs and increase the flow of blood in the leg veins.

This study will compare results from patients who receive the SCDs only to those who receive both SCD and anticoagulants. The outcome of this study will provide information about how best to prevent blood clots while not increase brain bleeding after head injury.

ELIGIBILITY:
Inclusion Criteria

The pragmatic nature of this study seeks to include all consecutive patients presenting with significant TBI, regardless of whether ICB is evident at presentation. Inclusion criteria are the following:

i) Patients with severe TBI defined as GCS of ≤8, or

ii) Patients with moderate TBI defined as GCS = 9-12, admitted to ICU, with at least some ICB present on initial CT scan and any of the following:

1. Requiring invasive mechanical ventilation at the time of screening
2. Increased ICB on repeat CT scan compared to initial CT scan

iii) Upon randomization the patient will be able to receive the first dose of study drug in the first 3 calendar days from the time of injury

iv) ≥ 18 years of age

Exclusion Criteria

All participants meeting any of the following exclusion criteria at baseline will be excluded from participation in this study:

i) Known Hypersensitivity to FRAGMIN (Dalteparin), or its constituents including benzyl alcohol or to other low molecular weight heparins and/or heparins or pork products

ii) Known history of confirmed or suspected immunologically-mediated heparin-induced thrombocytopenia (delayed-onset severe thrombocytopenia), and/or in patients with a known history of a positive in vitro platelet-aggregation test in the presence of FRAGMIN (Dalteparin) is positive

iii) Known septic endocarditis

iv) Uncontrollable active bleeding

v) Known major blood clotting disorders

vi) Known acute gastroduodenal ulcer (with active bleeding)

vii) Severe uncontrolled hypertension (i.e. BP>210 despite medications)

viii) Known diabetic or hemorrhagic retinopathy

ix) Anticipated to be unable to receive SCD on at least one lower extremity due to nature of injuries for duration of intervention period

x) Presence of another confounding factor that can adequately explain the poor GCS at time of presentation (e.g. drug toxicity, seizure)

xi) Known presence of irreversible coagulopathies

xii) Known Pregnancy

xiii) Participants extremely low weight (<45 kg), or extremely high weight (>120kg)

xiv) Not expected to survive more than 48 hours from admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2018-07-19 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Clinically important VTE | 8 days
  Composite outcome of clinically-important VTE within 7±1 days after randomization defined as any of:
  1. Symptomatic, objectively-confirmed pulmonary embolism (PE), or
  2. Symptomatic, objectively-confirmed, proximal leg deep vein thrombosis (DVT), or
  3. Proximal (above knee) leg DVT on compression ultrasonography on Day 7±1

SECONDARY OUTCOMES:
Clinically-important ICB (Intracranial bleeding) progression | 7 days
  Clinically-important ICB progression within 7±1 days after randomization , as defined by having (1) any increase in volume of blood in the brain on any CT scan within 7±1 days relative to initial CT scan on Day 0* AND (2) clinical worsening within 24 hours of this CT scan, defined by one or more of the following:
  * Surgical intervention related to increased ICB after Day 0 (craniotomy/craniectomy, ICP monitor, external ventricular drain)
  * Decrease of GCS (Glasgow Coma Scale) by at least 2 points not related to sedation
  * Increase in ICP >5 mmHg on 2 occasions at least 6 hours apart despite medical therapy (if ICP monitor is in place)
  * Death
Objectively confirmed new or progressing ICB on radiology, | 8 days
  Assessed by comparing the initial brain CT (Day 0) to that performed within 8±1 days following randomization (or most recent prior to death).
180-day Mortality | 180 days
  Mortality at 180 days
7-day Mortality | 7 days
  Mortality at 7 days
30-day Mortality | 30 days
  Mortality at 30 days
Delayed VTE after day 7 | 30 days
  Any clinically important VTE occurring between Day 8 to Day 30 detected by treating clinicians
Functional neurological outcome at day 30 as measured by Glasgow Outcome Scale Extended | 30 days
  Glasgow Outcome Scale Extended (GOSE) at Day 30±5 by phone interview.
Functional neurological outcome at day 180 as measured by Glasgow Outcome Scale Extended | 180 days
  Glasgow Outcome Scale Extended (GOSE) at Day 180±14 by phone interview.
Quality of life outcome at 30 days as measured by the EuroQol5D | 30 days
  EQ-5D (EuroQol 5D) at Day 30±5 by phone interview.
Quality of life outcome at 180 days as measured by the EuroQol5D | 180 days
  EQ-5D (EuroQol 5D) at Day 180±14 by phone interview.

CONTACTS AND LOCATIONS:
Overall Officials: Farhad Pirouzmand, MD, MSc, FRCSC, Principal Investigator — Sunnybrook Health Sciences Centre; Damon Scales, MD, PhD, FRCPC, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (12):
- Canada (12):
  - Foothills Medical Centre, Calgary, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Hamilton Health Sciences Centre, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Sunnybrook Health Science Centre, Toronto, Ontario
  - Unity Health Toronto, Toronto, Ontario
  - Hopital de L'Enfant-Jesus, Québec, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pirouzmand F, Mathieu F, Mansouri A, Kavikondala K, Alkins R, Boyd JG, Christie S, Couillard P, Cusimano MD, Engels PT, English S, Fourney D, Fowler R, Geerts W, Gooderham PA, Griesdale D, Hunter G, Jabehdar Maralani P, Kelly ME, Klein G, Kramer AH, Kromm J, Kutsogiannis DJ, Lauzier F, Machnowska M, Maslove DM, Mejia-Mantilla J, Midha R, Misra B, Murphy L, O'Kelly CJ, Patel C, Pinto RL, Pronovost AP, Sekhon M, Sharma SV, Sinclair J, Tsai E, Turgeon AF, Warade A, Scales DC; PROTEST investigators. Prophylaxis for venous thromboembolism in traumatic brain injury: protocol for a randomised controlled trial. BMJ Open. 2025 Dec 25;15(12):e114158. doi: 10.1136/bmjopen-2025-114158. PMID 41453781